CLINICAL TRIAL: NCT06945393
Title: EVALUATION OF THE EFFICACY OF ANTIPIGMENTING OR DEPIMENTING AGENTS UNDER PART OF VISIBLE LIGHT [400-450NM] EXPOSURES
Brief Title: ANTIPIGMENTING OR DEPIMENTING EFFICACY UNDER PART OF VISIBLE LIGHT
Acronym: ACR_BIOVI_21-0
Status: Completed | Type: Observational
Sponsor: L'Oreal (Industry)
Responsible Party: Sponsor
Other Study IDs: L'Oréal
Record Dates: First submitted 2025-04-18; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Visible Light Exposure on Healthy Back Skin
Keywords: pigmentation; visible light; antipigmentation; depigmentation
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 4 differents actives compare to its respective vehicle: 8 topical cosmetics formulae applied on the back of volunteers, in mini-zones about 9cm2, at 4mg/cm2. Applied twice daily during 46 days: T1: Kopcinol 5% in inverse silicon T2: Vitamin C 7% in inverse silicon T3: Thiopyridinone 1% in Bright Matte T4: CD7414 0.5% in Hydro Alcoholic gel T5: Vehicle Inverse silicon T6: Hydro Alcoholic gel vehicle T7: Bright Matte vehicle
  Interventions: Other: Cosmetic topical products

INTERVENTIONS:
Other: Cosmetic topical products — Cosmetic topical products efficacy evaluation

SUMMARY:
The study intends to validate a protocol and define a positive reference to evaluate the efficacy of anti-pigmenting and depigmenting agents under part of visible Light exposures, between 400nm to 450nm.

It is carried out on cosmetic products for which the safety has been assured by a toxicologist, with the aim of confirming the efficacy of the products, which will be used by a large number of consumers under normal and reasonably foreseeable use conditions.

DETAILED DESCRIPTION:
The main objective of this study is to assess the efficacy of antipigmenting or depigmenting agents under [400-450nm] exposure in healthy volunteers by skin colorimetry (Delta E).

The secondary objectives are:

* To assess the efficacy of antipigmenting or depigmenting agents under [400-450nm] exposure in healthy volunteers by clinical evaluation and additional colorimetry measurements (Delta L*, a*, b* and ITA°) and clinical evaluation.
* To assess the local tolerance and safety of the topical formulations under [400-450nm] exposure by recording adverse events and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy female or male volunteer from 18 to 50 years old
2. Skin type III-IV according to the Fitzpatrick classification
3. Average ITA° (Individual Typologic Angle calculated value) on the back between 18° and 32° at screening and inclusion visits with an allowed difference of ± 2° between screening and inclusion visits
4. Uniform skin color over the eight zones (difference in ITA° between each zone should not be more than 4°)
5. Absence of freckles, naevi, hypo or hyper pigmented regions, hairs and marks of bronzing on the investigational area on the back
6. Female subject of childbearing potential, who is not sexually active, or using an effective contraceptive method* for at least one month before the beginning of the study, and throughout the study or menopausal female (with absence of menstruations for less than one year) or post-menopausal female (with absence of menstruations for more than one year)
7. Female of childbearing potential or menopausal female (with absence of menstruations for less than one year) willing to undergo urine pregnancy test
8. Subject willing and able to fulfil the study requirements and schedule
9. Subject informed about the study objectives and procedures, and able to understand them
10. Subject who has given written inform consent

Exclusion Criteria:

1. Subject who is pregnant or lactating or who is planning to become pregnant during the study
2. Subject with BMI > 30
3. Having planned UV exposure of the investigational area (sunlight or sunbeds) throughout the study
4. Having used sunbeds or had excessive sun exposure of the investigational area within the 3 months before inclusion
5. Having sunburn (erythema) on the back
6. Dermatological disorders affecting the investigational area (presence of naevi, freckles, excess hair or uneven skin tones, vitiligo, photo-dermatological problems
7. History of skin cancer
8. History of abnormal response to sun
9. Presence of recent suntan (according to Investigator opinion) or photo-test marks
10. History of allergy, hypersensitivity, or any serious reaction to any cosmetic product
11. Any concomitant medical condition that may interfere with the study conduct in the opinion of the investigator
12. Having used within the month before inclusion any systemic medication for more than 5 consecutive days (e.g. steroidal and non-steroidal anti-inflammatory drugs, corticoids, insulin, antihistamines, antihypertensive, antibiotics such as quinolone, tetracycline, thiazides, fluoroquinolones)
13. Having used within the month before inclusion any medication known to cause abnormal responses to UV exposure (e.g. vitamin A derivative, psoralen, aminolevulinic acid derivatives, etc.), or having planned to use these medications during the study
14. Having used within the 3 months before inclusion any depigmenting / whitening or pro-pigmenting topical treatments, or any systemic treatment that would interfere with the study assessments (anti-inflammatory drugs, corticoids, retinoids, hydroquinone, etc.) or having planned to use these treatments during the study
15. Having used, within the past 6 months, any physical treatment including laser or phototherapy (PUVA, IPL, PDT…) on the investigational area, or having planned to use these treatments during the study
16. Having planned to perform intensive sport (> 5 hours per week) or swim during the study
17. Subject who declares to be deprived of freedom by administrative or legal decision
18. Subject who cannot be contacted by telephone in case of emergency
19. Subject having participated within the 30 days before inclusion or currently participating in another clinical study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy male and female volunteers from 18 to 50 yo, with Fitzpatrick III and IV and an ITA° between 18° to 32° at screening.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-10-21 (Actual); Primary Completion 2022-05-21 (Actual); Study Completion 2022-05-21 (Actual)

PRIMARY OUTCOMES:
Skin color measurement | from Day 1 to Day 47.
  Measurement of the skin color using Chromameter® (non-invasive assessment) between the exposed zone (ZE) and non-exposed zone (ZNE).

SECONDARY OUTCOMES:
Visual scoring of pigmentation | from Day 1 to Day 47.
  Visual evaluation of the pigmentation using L'Oreal pigmentation scale (0-13 points)
Visual scoring of erythema | from Day 1 to Day 47.
  Visual evaluation of the erythema using L'Oreal scale (0-13 points)

OTHER OUTCOMES:
Safety assessment | from Day 1 to Day 47.
  Safety will be assessed by recording Adverse Events, including cutaneous reactions (local intolerance), from the informed consent form signature date until the end of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- CIDP Roumania, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Piffaut V, De Dormael R, Belaidi JP, Bertrand L, Passeron T, Bernerd F, Marionnet C. Topical prevention from high energy visible light-induced pigmentation by 2-mercaptonicotinoyl glycine, but not by ascorbic acid antioxidant: 2 randomized controlled trials. Front Pharmacol. 2025 Oct 9;16:1651068. doi: 10.3389/fphar.2025.1651068. eCollection 2025. PMID 41142247